CLINICAL TRIAL: NCT03048708
Title: Changes in Thyroid Function Tests and Texture Following Bariatric Surgery Induced Weight Loss
Brief Title: Thyroid in Bariatric Surgery
Acronym: ThyrBar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Martin Weickert, Study Principal Investigator, University Hospitals Coventry and Warwickshire NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11/WM/0085; ID74554 (Other: IRAS)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Thyroid; Obesity; Insulin Resistance; Autoimmune Thyroiditis
Keywords: Bariatric surgery; Leptin; Thyroid function tests
MeSH Terms: conditions — Thyroid Diseases; Obesity; Insulin Resistance; Thyroiditis, Autoimmune | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese patients treated with bariatric surgery (Experimental): Patients with morbid obesity who were eligible for and willing to have bariatric surgery performed
  Interventions: Procedure: Bariatric surgery
- Obese patients not treated with bariatric surgery (No Intervention): Age and BMI matched patients with morbid obesity who either were not eligible for or were not willing to have bariatric surgery performed - no sufficient number of matched patients has completed the study; the arm of obese patients not treated with bariatric surgery has been discarded for the purpose of the analyses

INTERVENTIONS:
Procedure: Bariatric surgery — patients who had received treatment with bariatric surgery for medical reasons
  Arms: Obese patients treated with bariatric surgery

SUMMARY:
This study is expected to provide novel data regarding potential structural and functional changes of the thyroid gland in morbidly obese adults following significant weight loss through bariatric surgery. These data will complement evidence from epidemiological studies regarding the association of obesity and alterations in thyroid function. Potentially this study may justify further longer-term studies regarding the effects of weight gain and/or weight loss on the morphology of the thyroid gland and could help to form recommendations regarding follow-up investigations for the thyroid in morbidly obese patients.

DETAILED DESCRIPTION:
Alterations in thyroid function are reported in obesity. Thyroid hormones and thyroid-stimulating hormone (TSH) concentrations have been variously described as normal, elevated, or low in morbidly obese patients compared with normal weight controls. However, it is a common observation that a significant proportion of patients with morbid obesity display slightly increased serum levels of TSH, while even relatively mild elevations of serum TSH are associated with an increase in the occurrence of obesity. Of note, abnormalities in thyroid function and TSH mostly normalize after weight loss, suggesting that these biochemical alterations are reversible. Despite uncertainty regarding the underlying mechanisms, it has been suggested that neither autoimmunity nor iodine deficiency seems to play a critical role. Several alternative mechanisms leading to hyperthyrotropinemia have been hypothesized, which include impaired feedback due to decreased number of triiodothyronine (T3) receptors in the hypothalamus, and variations in peripheral deiodinase activity. Leptin, in addition to regulating body weight and satiation, has also been shown to mediate the production of pro-TRH in cultured fetal rat hypothalamic neurons. Partial regulation of TSH by leptin has been also reported in humans. In addition, peripheral thyroid hormone metabolism appears to be reflected by the ratio of T3 to reverse T3 (rT3) (T3/rT3-ratio). We have shown that the T3/rT3-ratio is significantly increased in insulin resistant patients compared to their insulin sensitive partners despite comparable TSH values. Given that obesity is strongly associated with insulin resistance, and thyroid hormones are known to modulate carbohydrate metabolism, e.g. by affecting cellular glucose uptake, possible changes in the T3/fT3 ratio following weight loss after bariatric surgery could be of interest.

Data from cross-sectional studies further indicate that the thyroid structure of obese patients can be also affected, independent of the existence of autoimmune thyroiditis as indicated by the presence of auto-antibodies such as TPO. Ultrasound (US) scans are able to accurately characterize the echographic structure of thyroid tissue, in addition to estimation of thyroid volume and identification of non-palpable thyroid nodules. The typical normal thyroid parenchyma has a distinct high echo density due to the follicle structure, which contrasts well with tissue of the collar muscles. The interface between thyroid cells and the colloid exhibits elevated acoustic impedance, causing high-frequency acoustic waves to be reflected back to the US probe. However, in autoimmune thyroid diseases both lymphocytic infiltration and disruption of normal tissue architecture cause a reduction in thyroid echogenicity, whereas other tissues close by such as muscle tissue appear to remain unaffected. Only few previous studies reported on the morphology of the thyroid gland in adults with morbid obesity. Given that thyroid function has been reported to return to normal after weight loss, research questions are also raised about the potential reversibility of thyroid structural abnormalities following substantial weight loss in previously morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Obesity (BMI > 40 kg/m2)
2. Age: 18-65

Exclusion Criteria:

1. Diagnosis of obesity secondary to primary endocrine or systemic disease (e.g. Cushing's syndrome)
2. Evidence of clinically relevant thyroid disease
3. Chronic systematic inflammatory disease (e.g. rheumatoid arthritis)
4. Pregnancy
5. Treatment with anti-inflammatory drugs (e.g. corticosteroids)
6. Type 1 diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in thyroid morphology and thyroid function tests in morbidly obese patients following significant weight loss after bariatric surgery | > 3 month or when relevant weight loss has been achieved
  Measurement of thyroid ultrasound (grey scale assessment, volume, echogenicity) and thyroid function tests (free T4, free T3, TSH and rT3) at baseline and at least 3 months after surgery when relevant weight loss is achieved

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho AHY, Ma SHX, Tan MKB, Bajpai RC. A Randomized Waitlist-Controlled Trial of an Intergenerational Arts and Heritage-Based Intervention in Singapore: Project ARTISAN. Front Psychol. 2021 Sep 6;12:730709. doi: 10.3389/fpsyg.2021.730709. eCollection 2021. PMID 34552538
- [Derived] Mapurunga MV, Andreoni S, de Oliveira DR, Sarubbi V Jr, Bonilha AC, D'Almeida V, Tomita L, Ramos LR, Demarzo M. Protocol for a Nested Randomized Controlled Trial to Evaluate the Feasibility and Preliminary Efficacy of the Mindfulness Based Health Promotion Program on the Quality of Life of Older Adults Assisted in Primary Care-"The MBHP-Elderly Study". Front Med (Lausanne). 2020 Nov 30;7:563099. doi: 10.3389/fmed.2020.563099. eCollection 2020. PMID 33425931
- [Derived] Beit Yosef A, Jacobs JM, Shenkar S, Shames J, Schwartz I, Doryon Y, Naveh Y, Khalailh F, Berrous S, Gilboa Y. Activity Performance, Participation, and Quality of Life Among Adults in the Chronic Stage After Acquired Brain Injury-The Feasibility of an Occupation-Based Telerehabilitation Intervention. Front Neurol. 2019 Dec 6;10:1247. doi: 10.3389/fneur.2019.01247. eCollection 2019. PMID 31866924
- [Derived] Kyrou I, Adesanya O, Hedley N, Wayte S, Grammatopoulos D, Thomas CL, Weedall A, Sivaraman S, Pelluri L, Barber TM, Menon V, Randeva HS, Tedla M, Weickert MO. Improved Thyroid Hypoechogenicity Following Bariatric-Induced Weight Loss in Euthyroid Adults With Severe Obesity-a Pilot Study. Front Endocrinol (Lausanne). 2018 Aug 24;9:488. doi: 10.3389/fendo.2018.00488. eCollection 2018. PMID 30197625